CLINICAL TRIAL: NCT05484518
Title: Is Method of Levels (MOL) an Acceptable and Feasible Psychological Intervention for People Using Community Based Crisis Services? A Case Series.
Brief Title: Method of Levels for People Using Community Crisis Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Sara Goodier, Student/Chief Investigator, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 316034
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2022-12

CONDITIONS: Individuals Presenting to Crisis Services

STUDY DESIGN:
Intervention Model Description: Case series
Masking Description: One group only, no masking required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Method of Levels Therapy (Experimental): Method of levels therapy, see intervention details. All participants will receive therapy and must attend a minimum of one session for their data to be included in the study.
  Interventions: Behavioral: Method of Levels Therapy

INTERVENTIONS:
Behavioral: Method of Levels Therapy — Method of Levels (MOL) is a therapy that is the direct application of Perceptual Control Theory (PCT) (Powers, 2008) which proposes that psychological distress results from a person's reduced control over important life goals. A conflict between two or more goals can occur outside of a person's awareness (Carey, Mansell & Tai, 2014) and the achievement of one goal leaves the other incompatible goal unachievable, leading to distress (Mansell, 2012). MOL therapy aims to help people develop awareness of important goals and conflicts between them, to increase their chances of developing potential solutions. Conflict can be resolved through reorganisation; a mechanism through which random change is continuously generated until control is restored (Tai, 2016).
  Therapy uses a questioning style to help clients bring their attention to their problems long enough for them to restore control. In practice clients choose the number, frequency and duration of therapy sessions

SUMMARY:
A mental health crisis is when someone is so distressed they need urgent help from services; often because they behave in ways that poses risk to themselves or others. Crisis teams offer care in the community to support people at home rather than in hospital. Current psychological interventions offered by crisis teams tend to be short-term and mainly involve providing information about the difficulties people are experiencing and help them to develop skills, such people as problem solving. This can be useful, however providing more intensive psychological support has been much more difficult within crisis settings, as teams must use limited resources to focus on managing risk. A therapy, called Method of Levels (MOL), designed to be flexible, may be helpful to add to treatment offered by crisis services in the community.

MOL aims to help people hold their attention on a problem long enough to view it in different ways, so that they might think of new solutions. This works by helping a person to regain a sense of control in their life and feel less distressed. MOL is useful for working with lots of different issues, since therapy does not only focus on one type of problem. People also get to choose what is discussed in therapy and session structure.

Research has shown MOL can be useful for people in crisis in places such as inpatient settings. So far, no research has been conducted within the community for people in crisis. This study aims to examine if MOL can be delivered within a crisis service in a way that is helpful and acceptable to people. To do this, the investigators will offer MOL to a small number of people presenting to crisis teams and collect information on whether people take up the therapy, and their experience of receiving it.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged over 18 years.
2. Meet criteria for crisis services and currently working with the crisis team
3. Able to provide informed consent (no queries regarding capacity)
4. Willing to engage in psychological therapy.
5. Ability to speak English fluently enough to provide informed consent and engage in therapy.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Inability to speak English fluently enough to engage in therapy: As MOL is a therapy that relies on mobilising attention, the use of interpreters during therapy for non-English speakers may serve to alter the participants attention differently. This may confound results; as this is a preliminary case series, it would not be appropriate to include non-English speakers.
3. Problems of an organic nature, or a learning disability that might affect cognitive functioning.
4. Substance misuse as primary presenting problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate. | Length of study (up to one year)
  Number of participants recruited into the study.
Retention rate. | Length of study (up to one year)
  Number of participants retained to the end of the study.
Psychological Outcome Profiles. | Beginning of each therapy session for length of therapy (chosen by participant), up to 5 months
  Quantitative measure to indicate acceptability. Total score between 0-20, where a lower score indicates a better outcome.
Session Rating Scale. | End of each therapy session (chosen by participant), up to 5 months.
  Quantitative measure to indicate acceptability.Total score between 0-40, where a lower score indicates a better outcome.
Qualitative interviews | End of therapy, up to 5 months.
  Thematic analysis of qualitative interviews following end of therapy.

SECONDARY OUTCOMES:
Clinical Outcomes in Routine Evaluation Outcome Measure | On recruitment, monthly (up to 5 months), one month follow up
  Questionnaire. Total score between 0-136, where a lower score indicates a better outcome.
Reorganisation of Conflict Scale. | On recruitment, monthly (up to 5 months), one month follow up
  Questionnaire. 22 self reported items, each on a scale of 0-100, where a lower score indicates a better outcome.
Suicidal ideation Attributes Scale. | On recruitment, monthly (up to 5 months), one month follow up
  Questionnaire. Total score of 0-50, where a higher score indicates more severe suicidal thoguhts.
BBC Subjective Well-being scale (BBC-SWB) (Kinderman, Schwannauer, Pontin, & Tai, 2011). | On recruitment, monthly (up to 5 months), one month follow up
  Questionnaire. 24 items scores on a 5 point likert scale, where 5 indiicates high wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Goodier, MSc, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No